CLINICAL TRIAL: NCT01961037
Title: Translation of an Evidence-Based Fall-Prevention Program Into Rural West Virginia Churches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dina L Jones, PT, PhD, Associate Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5 R49 CE002109-DLJ; 5R49CE002109 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-10-11 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Tai Chi; Older Adults; Balance; Moving for Better Balance; Church; Congregational Intervention; Rural; West Virginia
MeSH Terms: interventions — Tai Ji; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity intervention (Experimental): Tai Chi: Moving for Better Balance exercise program
  Interventions: Other: Tai Chi: Moving for Better Balance

INTERVENTIONS:
Other: Tai Chi: Moving for Better Balance — Participants will attend one-hour Tai Chi classes twice weekly for 16 weeks.
  Other Names: Tai Chi; Exercise; Physical Activity

SUMMARY:
Falls are the leading cause of death and injuries in adults over age 65 both nationally and in West Virginia. Rurality, age, physical inactivity, and chronic conditions, such as arthritis, are strong risk factors for falls in this population. West Virginia has a higher than average fall rate, the second oldest population, the greatest proportion of inactive adults, and the second highest prevalence of arthritis in the US. Thus, older adults in rural West Virginia are at high risk for falls and in great need of public health fall prevention programs. The Tai Chi: Moving for Better Balance (MFBB) program is a community-based, fall-prevention exercise program for older adults. A waiver of informed consent will be requested to conduct the telephone screenings to determine study eligibility. We will enroll up to 300 people in classes to be held at 20 churches in West Virginia. Classes will be held twice per week for 16 weeks and taught by certified MFBB instructors. Participants will be interviewed by telephone, have a brief physical function ability exam, and complete a questionnaire before starting the exercise class, at the end of the class, and 4 months later. The study is being conducted to answer the following questions: 1) What are the functional improvements of older adults who participate in a 16-week MFBB program; 2) What is the rate of falls for those adults; 3) What is the rate and severity of those fall-related injuries of the MFBB participants? The purpose of the study is to: 1) implement a 16-week intervention of MFBB with a 16-week follow-up, in older adults in churches in rural West Virginia; 2) describe functional and fall/injury outcomes. Ultimately, we will translate an efficacious and effective fall-prevention intervention into a new setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or older

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
10-Meter Walk Test | 16 weeks
  A timed 10-Meter Walk Test at a self-selected walking speed will be used to determine gait speed

SECONDARY OUTCOMES:
Number of fall-related injuries | 32 weeks
  Measure the number of reported fall-related injuries by study participants during the intervention and during the 16-week period after the intervention is complete.
Number of falls | 32 weeks
  Measure the number of reported falls by study participants during the intervention and during the 16-week period after the intervention is complete.

OTHER OUTCOMES:
Four Square Test | 16 weeks
  Balance will be assessed using the Four Square Test which requires participants to step over low objects and move in four directions.
Timed Up-And-Go Test | 16 weeks
  The Timed Up-And-Go Test will be used to assess functional mobility. A participant stands from a chair, walks three meters at a self-selected pace, turns, and returns to the chair to sit.
Champs Activity Questionnaire for Older Adults | 16 weeks
  The CHAMPS Activities Questionnaire for Older Adults will be administered by telephone interview by trained team members to assess the typical weekly frequency and duration of participation in 41 leisure and daily activities during the past month. The CHAMPS has shown superior reliability, validity, and responsiveness over other instruments in trials of fall-injury prevention programs.
SF-12 | 16 weeks
  The SF-12 v2, which is recommended for inclusion in fall/injury prevention trials, will be used to determine physical and mental health-related quality of life.
Falls Efficacy Scale | 16 weeks
  The 10-item reliable and valid Falls Efficacy Scale will be utilized to assess fear of falling.
Translation of MFBB in the churches with respect to its Reach | 16 weeks
  We will determine the proportion of eligible older adults who participate in a 16-week church-based intervention of MFBB.
Translation of MFBB in the churches with respect to its Adoption | 16 weeks
  We will determine the proportion of invited churches that offer MFBB.
Translation of MFBB in the churches with respect to its Implementation | 16 weeks
  We will determine if MFBB was delivered as intended by its developer.
Translation of MFBB in the churches with respect to its Maintenance (churches) | 32 weeks
  We will determine the proportion of churches who continue MFBB at 32 weeks.
Translation of MFBB in the churches with respect to its Maintenance (participants) | 32 weeks
  We will determine the proportion of participants who continue MFBB at 32 weeks.
10-Meter Walk Test | 32 weeks
  A timed 10-Meter Walk Test at a self-selected walking speed will be used to determine gait speed.
Four Square Test | 32 weeks
  Balance will be assessed using the Four Square Test which requires participants to step over low objects and move in four directions.
Timed Up-And-Go Test | 32 weeks
  The Timed Up-And-Go Test will be used to assess functional mobility. A participant stands from a chair, walks three meters at a self-selected pace, turns, and returns to the chair to sit.
Champs Activity Questionnaire for Older Adults | 32 weeks
  The CHAMPS Activities Questionnaire for Older Adults will be administered by telephone interview by trained team members to assess the typical weekly frequency and duration of participation in 41 leisure and daily activities during the past month. The CHAMPS has shown superior reliability, validity, and responsiveness over other instruments in trials of fall-injury prevention programs.
SF-12 | 32 weeks
  The SF-12 v2, which is recommended for inclusion in fall/injury prevention trials, will be used to determine physical and mental health-related quality of life.
Falls Efficacy Scale | 32 weeks
  The 10-item reliable and valid Falls Efficacy Scale will be utilized to assess fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Dina L Jones, PT, PhD, Principal Investigator — West Virginia University
Locations (9):
- United States (9):
  - Hughes River Presbyterian Church, Cairo, West Virginia
  - Wesley United Methodist Church, Ellenboro, West Virginia
  - Harper Memorial Church, Gandeeville, West Virginia
  - First Baptist Church, Grantsville, West Virginia
  - First Assembly of God, Harrisville, West Virginia
  - Cisco Community Church, Petroleum, West Virginia
  - First Baptist Church, Spencer, West Virginia
  - Memorial United Methodist Church, Spencer, West Virginia
  - Spencer Presbyterian Church, Spencer, West Virginia